CLINICAL TRIAL: NCT01525628
Title: A Multi-centre, Open Label, Parallel Group Trial to Evaluate the Pharmacokinetic Interactions Between BI 207127 (600 mg t.i.d. or 600 mg b.i.d.) and BI 201335 (120 mg q.d.) Given in Combination With Ribavirin for 24 Weeks, and Their Combined Effect on the Pharmacokinetics of Tenofovir, Raltegravir, Caffeine (the Probe Drug Substrate for CYP1A2), Tolbutamide (the Probe Drug Substrate for CYP2C9) and Midazolam (the Probe Drug Substrate for CYP3A4) in Treatment naïve Patients and Prior Treatment Relapse or Partial Responder Patients With Genotype 1 Chronic Hepatitis C Infection
Brief Title: Drug Drug Interaction Study Between BI 201335 and BI 207127 in Chronic Hepatitis C Infected Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1241.27; 2012-004102-10 (EudraCT Number: EudraCT)
Record Dates: First submitted 2012-02-01; First posted 2012-02-03 (Estimated); Results first posted 2016-06-10 (Estimated); Last update posted 2016-06-10 (Estimated); Status verified 2016-05

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Midazolam; faldaprevir; Tenofovir; Caffeine; Tolbutamide; deleobuvir; Ribavirin

ARMS (5):
- Group A (Experimental): Effect of BI 207127 on BI 201335, the effect of BI 201335 and dual oral direct acting antiviral (DAAs) on caffeine, tolbutamide and midazolam
  Interventions: Drug: tolbutamide; Drug: midazolam; Drug: caffeine; Drug: BI 201335; Drug: pegylated interferon; Drug: BI 207127; Drug: ribavirin
- Group B (Experimental): Effect of BI 201335 on BI 207127, the effect of BI 207127 and metabolites and dual oral DAAs on caffeine, tolbutamide and midazolam
  Interventions: Drug: BI 201335; Drug: caffeine; Drug: tolbutamide; Drug: pegylated interferon; Drug: BI 207127; Drug: ribavirin; Drug: midazolam
- Group C (Experimental): Effect of Dual oral DAAs on tenofovir
  Interventions: Drug: tenofovir; Drug: BI 207127; Drug: ribavirin; Drug: BI 201335
- Group D (Experimental): Effect of BI 201335 and BI 207127 at 600 mg b.i.d. on caffeine, tolbutamide and midazolam
  Interventions: Drug: midazolam; Drug: BI 201335; Drug: BI 207127; Drug: ribavirin; Drug: caffeine; Drug: tolbutamide
- Group E (Experimental): Effect of BI 201335 and BI 207127 on raltegravir
  Interventions: Drug: BI 201335; Drug: ribavirin; Drug: BI 207127

INTERVENTIONS:
Drug: midazolam — CYP3A probe drug
  Arms: Group D
Drug: BI 201335 — HCV protease inhibitor
  Arms: Group B
Drug: tenofovir — nucleoside analogue
  Arms: Group C
Drug: caffeine — CYP1A2 probe drug
  Arms: Group B
Drug: tolbutamide — CYP2C9 probe drug
  Arms: Group B
Drug: tolbutamide — CYP2C9 probe drug
  Arms: Group A
Drug: midazolam — CYP3A probe drug
  Arms: Group A
Drug: caffeine — CYP1A2 probe drug
  Arms: Group A
Drug: pegylated interferon — HCV treatment
  Arms: Group B
Drug: BI 201335 — HCV protease inhibitor
  Arms: Group D
Drug: BI 201335 — HCV protease inhibitor
  Arms: Group E
Drug: BI 207127 — HCV polymerase inhibitor
  Arms: Group C
Drug: BI 207127 — HCV polymerase inhibitor
  Arms: Group D
Drug: BI 201335 — HCV protease inhibitor
  Arms: Group A
Drug: BI 207127 — HCV polymerase inhibitor
  Arms: Group B
Drug: ribavirin — HCV treatment
  Arms: Group B
Drug: ribavirin — HCV treatment
  Arms: Group C
Drug: ribavirin — HCV treatment
  Arms: Group E
Drug: pegylated interferon — HCV treatment
  Arms: Group A
Drug: ribavirin — HCV treatment
  Arms: Group D
Drug: caffeine — CYP1A2 probe drug
  Arms: Group D
Drug: tolbutamide — CYP2C9 probe drug
  Arms: Group D
Drug: BI 207127 — HCV polymerase inhibitor
  Arms: Group A
Drug: midazolam — CYP3A probe drug
  Arms: Group B
Drug: BI 201335 — HCV protease inhibitor
  Arms: Group C
Drug: BI 207127 — HCV polymerase inhibitor
  Arms: Group E
Drug: ribavirin — HCV treatment
  Arms: Group A

SUMMARY:
To evaluate the drug-drug interactions between BI 201335 and BI 207127 as well as their combined effect on CYP probe drug substrates and on tenofovir and raltegravir in treatment naive or prior treatment relapse patients with chronic hepatitis C infection.

ELIGIBILITY:
Inclusion criteria:

1. Chronic hepatitis C genotype 1 infection, diagnosed at least 6 months prior to screening
2. Treatment naive or confirmed prior treatment relapse or partial response following treatment with interferon and ribavirin
3. Age 18 to 70 years
4. HCV RNA (Hepatitis C Virus RiboNucleic Acid) = 1,000 IU/mL at screening
5. Liver biopsy or fibroscan to exclude cirrhosis

Exclusion criteria:

1. Hepatitis C Virus (HCV) infection of mixed genotype; Hepatitis B Virus (HBV) or Human Immunodeficiency Virus (HIV) co-infection
2. Evidence of acute or chronic liver disease due to causes other than chronic HCV infection,
3. Decompensated liver disease, or history of decompensated liver disease,
4. Body weight < 40 or > 125 kg,
5. Clinical evidence of significant or unstable cardiovascular disease, chronic pulmonary disease, history or evidence of retinopathy or clinically significant ophthalmological disorder
6. Pre-existing psychiatric condition that could interfere with the subject's participation in and completion of the study
7. Laboratory parameters disorders (thalassemia major, sickle cell anemia or glucose 6 phosphate dehydrogenase deficit)
8. Hemoglobin < 12 g/dL for women and < 13 g/dL for men
9. Patients who have been previously treated with at least one dose of any antiviral or immunomodulatory drug other than interferon alfa or ribavirin for acute or chronic HCV infection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2012-04; Primary Completion 2013-12 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (16):
- United States (5):
  - 1241.27.0006 Boehringer Ingelheim Investigational Site, La Mesa, California
  - 1241.27.0005 Boehringer Ingelheim Investigational Site, Rockville, Maryland
  - 1241.27.0004 Boehringer Ingelheim Investigational Site, Marlton, New Jersey
  - 1241.27.0003 Boehringer Ingelheim Investigational Site, Philadelphia, Pennsylvania
  - 1241.27.0001 Boehringer Ingelheim Investigational Site, Salt Lake City, Utah
- Canada (7):
  - 1241.27.0200 Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - 1241.27.0600 Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - 1241.27.0700 Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - 1241.27.0400 Boehringer Ingelheim Investigational Site, Victoria, British Columbia
  - 1241.27.0100 Boehringer Ingelheim Investigational Site, London, Ontario
  - 1241.27.0300 Boehringer Ingelheim Investigational Site, Ottawa, Ontario
  - 1241.27.0500 Boehringer Ingelheim Investigational Site, Montreal, Quebec
- Germany (4):
  - 1241.27.4907 Boehringer Ingelheim Investigational Site, Cologne
  - 1241.27.4901 Boehringer Ingelheim Investigational Site, Frankfurt am Main
  - 1241.27.4903 Boehringer Ingelheim Investigational Site, Leipzig
  - 1241.27.4906 Boehringer Ingelheim Investigational Site, Mainz

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 72 patients were treated and analysed.
Pre-assignment Details: This was randomised (Groups A and B only), controlled, open-label, parallel-group (Groups A to E), multi-centre trial in treatment-naive patients and patients with prior treatment relapse or partial responders with Genotype 1 (GT1) chronic Hepatitis C infection.
Groups:
- Group A: 600mg deleobuvir(DBV) tablet taken orally 3 times a day plus 120mg faldaprevir(FDV) capsule taken orally once daily plus ribavirin(RBV) tablet taken orally twice daily for 24 weeks along with pegylated interferon α-2a(PegIFN) injection and probe drugs(200 mg caffeine tablet, 500 mg tolbutamide tablet, and 2 mg midazolam syrup administered orally on days 1, 9, 17, and 66). In group A the effect of DBV on FDV, the effect of FDV, dual oral direct acting antiviral (DAAs) and their metabolites on caffeine, tolbutamide and midazolam were determined.
- Group B: 600mg deleobuvir(DBV) tablet taken orally 3 times a day plus 120mg faldaprevir(FDV) capsule taken orally once daily plus ribavirin(RBV) tablet taken orally twice daily for 24 weeks along with pegylated interferon α-2a (PegIFN) injection and probe drugs(200 mg caffeine tablet, 500 mg tolbutamide tablet, and 2 mg midazolam syrup administered orally on days 1, 9, 17, and 66). In group B the effect of FDV on DBV, the effect of DBV, dual oral direct acting antiviral (DAAs) and their metabolites on caffeine, tolbutamide and midazolam were determined.
- Group C: 600mg deleobuvir(DBV) tablet taken twice a day plus 120mg faldaprevir(FDV) capsule taken orally once daily plus ribavirin(RBV) tablet taken orally twice daily for 24 weeks with tenofovir tablet 300mg daily on days 1-17.
- Group D: 600mg deleobuvir(DBV) tablet taken twice a day plus 120mg faldaprevir(FDV) capsule taken orally once daily plus ribavirin(RBV) tablet taken orally twice daily with probe drugs(200 mg caffeine tablet, 500 mg tolbutamide tablet, and 2 mg midazolam syrup administered orally on days 1, 9, 17, and 66).
- Group E: 600mg deleobuvir(DBV) tablet taken twice a day plus 120mg faldaprevir(FDV) capsule taken orally once daily plus ribavirin(RBV) tablet taken orally twice daily for 24 weeks with raltegravir tablet 400mg twice daily on days 1-17.
Period: Overall Study
Arm/Group | Group A | Group B | Group C | Group D | Group E
Started | 16 | 19 | 16 | 14 | 7
Completed | 14 | 14 | 11 | 10 | 4
Not Completed | 2 | 5 | 5 | 4 | 3
Not completed — Adverse Event | 1 | 1 | 2 | 0 | 1
Not completed — Lack of Efficacy | 0 | 2 | 2 | 1 | 2
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0
Not completed — Other reason not defined above | 0 | 0 | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Population: The treated set (TRT) included all patients who were dispensed trial medication and were documented to have taken at least one dose of trial drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Group C | Group D | Group E | Total
Number analyzed (Participants) | 16 | 19 | 16 | 14 | 7 | 72
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.2 (12.3) | 53.6 (9.3) | 53.1 (9.5) | 48.4 (12.7) | 52.1 (10.4) | 51.1 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 5 | 7 | 1 | 28
  Male | 9 | 11 | 11 | 7 | 6 | 44

OUTCOME MEASURES:

1. Primary Outcome: Cmax of Faldaprevir (BI 201335)
Description: Maximum concentration of an analyte in plasma
Time Frame: PK plasma samples were taken at: 5 minutes before drug administration and 1 hour (h), 2h, 3h, 4h, 5h, 5:55h, 8h, 10h, 11:55h, 15h, 23:55h after first drug administration on days 9, 17 and 66.
Population: The pharmacokinetic set (PKS): included all patients in the treated set who provided at least one observation for at least one primary (PK) endpoint without important protocol violations relevant to the evaluation of PK. This endpoint was not planned to be analysed for groups C, D and E.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Group A | Group B
Number analyzed (Participants) | 16 | 19
ng/mL
  Day 9 (N=15,0) | 3520 (54.8) | NA (NA) — Not calculated as this timepoint was not planned to be analysed for group B.
  Day 17 (N=14,14) | 8780 (47.5) | 9950 (51.0)
  Day 66 (N=13,15) | 4410 (48.7) | 6690 (78.8)
Statistical Analysis 1: Comparison: Group A; Day 17 vs. Day 9; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 1.0000, ANOVA; ANOVA (analysis of variance) model on the logarithm scale was used with 'subject' as random, whereas the 'treatment' as fixed effect; Ratio of gmeans Day 17 vs. Day 9 (%) = 251.37, 90% CI 2-sided [205.54 to 307.43], Standard Deviation 31.0 — Relative bioavailability of BI 201335 at Day 17 vs. Day 9 -was estimated by the ratios of the adjusted geometric means (gMean). Standard deviation is actually Intra individual geometric coefficient variation (gCV)
Statistical Analysis 2: Comparison: Group A; Day 66 vs. Day 9; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 0.6514, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 66 vs. Day 9 (%) = 131.30, 90% CI 2-sided [105.40 to 163.57], Standard Deviation 32.5 — Relative bioavailability of BI 201335 at Day 66 vs. Day 9 -was estimated by the ratios of the adjusted geometric means (gMean). Standard deviation is actually Intra individual geometric coefficient variation (gCV)

2. Primary Outcome: C24hr of Faldaprevir (BI 201335)
Description: Concentration of an analyte in plasma at 24 hours
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Group A | Group B
Number analyzed (Participants) | 16 | 19
ng/mL
  Day 9 (N=15,0) | 983 (65.5) | NA (NA) — Not calculated as this timepoint was not planned to be analysed for group B.
  Day 17 (N=14,19) | 3670 (90.4) | 5410 (91.6)
  Day 66 (N=13,14) | 1140 (107) | 2580 (135)
Statistical Analysis 1: Comparison: Group A; Day 17 vs. Day 9; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 1.0000, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 17 vs. Day 9 (%) = 381.11, 90% CI 2-sided [317.01 to 458.19], Standard Deviation 28.1 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Group A; Day 66 vs. Day 9; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 0.4718, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 66 vs. Day 9 (%) = 123.65, 90% CI 2-sided [94.66 to 161.51], Standard Deviation 40.0 — [estimate comment as in outcome 1, analysis 2]

3. Primary Outcome: Area Under the Concentration-time Curve (AUC) of Faldaprevir (BI 201335) From 0 to 24 Hours
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to 24 hours
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Group A | Group B
Number analyzed (Participants) | 16 | 19
ng*h/mL
  Day 9 (N=15,0) | 45600 (54.5) | NA (NA) — Not calculated as this timepoint was not planned to be analysed for group B.
  Day 17 (N=14,19) | 138000 (62.1) | 173000 (60.8)
  Day 66 (N=13,15) | 56200 (58.2) | 97300 (114)
Statistical Analysis 1: Comparison: Group A; Day 17 vs. Day 9; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 1.0000, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 17 vs. Day 9 (%) = 306.45, 90% CI 2-sided [250.93 to 374.26], Standard Deviation 30.7 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Group A; Day 66 vs. Day 9; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 0.6185, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 66 vs. Day 9 (%) = 129.85, 90% CI 2-sided [104.26 to 161.71], Standard Deviation 32.5 — [estimate comment as in outcome 1, analysis 2]

4. Primary Outcome: Cmax of Deleobuvir (BI 207127)
Description: Maximum concentration of an analyte in plasma
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Group A | Group B
Number analyzed (Participants) | 16 | 19
nmol/L
  Day 9 (N=0, 17) | NA (NA) — Not calculated as this timepoint was not planned to be analysed for group A. | 10900 (85.3)
  Day 17 (N=14, 19) | 27000 (64.6) | 31400 (45.8)
  Day 66 (N=13, 15) | 10100 (78.2) | 16000 (100)
Statistical Analysis 1: Comparison: Group B; Day 17 vs. Day 9; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 1.0000, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 17 vs. Day 9 (%) = 286.01, 90% CI 2-sided [228.51 to 357.97], Standard Deviation 39.4 — Relative bioavailability of BI 207127 at Day 17 vs. Day 9 -was estimated by the ratios of the adjusted geometric means (gMean). Standard deviation is actually Intra individual geometric coefficient variation (gCV)
Statistical Analysis 2: Comparison: Group B; Day 66 vs. Day 9; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 0.8210, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 66 vs. Day 9 (%) = 150.45, 90% CI 2-sided [106.81 to 211.91], Standard Deviation 55.1 — Relative bioavailability of BI 207127 at Day 66 vs. Day 9 -was estimated by the ratios of the adjusted geometric means (gMean). Standard deviation is actually Intra individual geometric coefficient variation (gCV)

5. Primary Outcome: C6hr of Deleobuvir (BI 207127)
Description: Concentration of an analyte in plasma at 6 hours
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Group A | Group B
Number analyzed (Participants) | 16 | 19
nmol/L
  Day 9 (N=0, 17) | NA (NA) — Not calculated as this timepoint was not planned to be analysed for group A. | 5800 (129)
  Day 17 (N=14, 19) | 17900 (84.2) | 20800 (83.8)
  Day 66 (N=13, 14) | 5080 (108) | 10100 (133)
Statistical Analysis 1: Comparison: Group B; Day 17 vs. Day 9; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 1.0000, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 17 vs. Day 9 (%) = 349.90, 90% CI 2-sided [269.12 to 454.93], Standard Deviation 46.4 — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Group B; Day 66 vs. Day 9; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 0.9533, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 66 vs. Day 9 (%) = 176.56, 90% CI 2-sided [125.95 to 247.50], Standard Deviation 50.1 — [estimate comment as in outcome 4, analysis 2]

6. Primary Outcome: AUC 0-6hr of Deleobuvir (BI 207127)
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to 6 hours
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | Group A | Group B
Number analyzed (Participants) | 16 | 19
nmol*h/L
  Day 9 (N=0, 17) | NA (NA) — Not calculated as this timepoint was not planned to be analysed for group A. | 41100 (93.7)
  Day 17 (N=14, 19) | 119000 (73.7) | 135000 (65.0)
  Day 66 (N=13, 15) | 36200 (89.0) | 59200 (129)
Statistical Analysis 1: Comparison: Group B; Day 17 vs. Day 9; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 1.0000, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 17 vs. Day 9 (%) = 322.68, 90% CI 2-sided [256.24 to 406.34], Standard Deviation 40.4 — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Group B; Day 66 vs. Day 9; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 0.7461, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 66 vs. Day 9 (%) = 145.93, 90% CI 2-sided [97.83 to 217.69], Standard Deviation 66.2 — [estimate comment as in outcome 4, analysis 2]

7. Primary Outcome: Cmax of Deleobuvir Metabolite Acyl-glucuronide (BI 208333)
Description: Maximum concentration of an analyte in plasma
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Group A | Group B
Number analyzed (Participants) | 16 | 19
nmol/L
  Day 9 (N=0, 17) | NA (NA) — Not calculated as this timepoint was not planned to be analysed for group A. | 5620 (119)
  Day 17 (N=14, 19) | 12700 (89.4) | 20200 (111)
  Day 66 (N=13, 15) | 3790 (66.9) | 6550 (98.3)
Statistical Analysis 1: Comparison: Group B; Day 17 vs. Day 9; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 1.0000, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 17 vs. Day 9 (%) = 355.04, 90% CI 2-sided [298.13 to 422.83], Standard Deviation 29.9 — Relative bioavailability of BI 208833 at Day 17 vs. Day 9 -was estimated by the ratios of the adjusted geometric means (gMean). Standard deviation is actually Intra individual geometric coefficient variation (gCV)
Statistical Analysis 2: Comparison: Group B; Day 66 vs. Day 9; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 0.4337, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 66 vs. Day 9 (%) = 120.67, 90% CI 2-sided [83.68 to 174.01], Standard Deviation 58.3 — Relative bioavailability of BI 208833 at Day 66 vs. Day 9 -was estimated by the ratios of the adjusted geometric means (gMean). Standard deviation is actually Intra individual geometric coefficient variation (gCV)

8. Primary Outcome: C6hr of Deleobuvir Metabolite Acyl-glucuronide (BI 208333)
Description: Concentration of an analyte in plasma at 6 hours
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Group A | Group B
Number analyzed (Participants) | 16 | 19
nmol/L
  Day 9 (N=0, 17) | NA (NA) — Not calculated as this timepoint was not planned to be analysed for group A. | 4330 (154)
  Day 17 (N=14, 19) | 11200 (83.7) | 17500 (119)
  Day 66 (N=13, 14) | 2740 (85.9) | 5780 (132)
Statistical Analysis 1: Comparison: Group B; Day 17 vs. Day 9; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 1.0000, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 17 vs. Day 9 (%) = 397.73, 90% CI 2-sided [330.79 to 478.22], Standard Deviation 31.6 — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 2: Comparison: Group B; Day 66 vs. Day 9; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 0.7346, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 66 vs. Day 9 (%) = 142.27, 90% CI 2-sided [99.49 to 203.44], Standard Deviation 53.1 — [estimate comment as in outcome 7, analysis 2]

9. Primary Outcome: AUC 0-6hr of Deleobuvir Metabolite Acyl-glucuronide (BI 208333)
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to 6 hours
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | Group A | Group B
Number analyzed (Participants) | 16 | 19
nmol*h/L
  Day 9 (N=0, 17) | NA (NA) — Not calculated as this timepoint was not planned to be analysed for group A. | 24300 (131)
  Day 17 (N=14, 19) | 61800 (97.9) | 98800 (124)
  Day 66 (N=13, 15) | 15000 (81.2) | 27600 (128)
Statistical Analysis 1: Comparison: Group B; Day 17 vs. Day 9; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 1.0000, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 17 vs. Day 9 (%) = 403.86, 90% CI 2-sided [332.19 to 490.99], Standard Deviation 33.6 — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 2: Comparison: Group B; Day 66 vs. Day 9; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 0.3968, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 66 vs. Day 9 (%) = 116.96, 90% CI 2-sided [75.38 to 181.47], Standard Deviation 73.1 — [estimate comment as in outcome 7, analysis 2]

10. Primary Outcome: Cmax of Deleobuvir Reduction Metabolite CD 6168
Description: Maximum concentration of an analyte in plasma
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Group A | Group B
Number analyzed (Participants) | 16 | 19
nmol/L
  Day 9 (N=0, 17) | NA (NA) — Not calculated as this timepoint was not planned to be analysed for group A. | 3040 (115)
  Day 17 (N=14, 19) | 8520 (119) | 12400 (70.9)
  Day 66 (N=13, 15) | 4510 (117) | 8880 (111)
Statistical Analysis 1: Comparison: Group B; Day 17 vs. Day 9; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 1.0000, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 17 vs. Day 9 (%) = 408.66, 90% CI 2-sided [315.15 to 529.90], Standard Deviation 45.9 — Relative bioavailability of BI CD 6168 at Day 17 vs. Day 9 -was estimated by the ratios of the adjusted geometric means (gMean). Standard deviation is actually Intra individual geometric coefficient variation (gCV)
Statistical Analysis 2: Comparison: Group B; Day 66 vs. Day 9; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 0.9993, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 66 vs. Day 9 (%) = 301.19, 90% CI 2-sided [204.61 to 443.35], Standard Deviation 62.1 — Relative bioavailability of BI CD 6168 at Day 66 vs. Day 9 -was estimated by the ratios of the adjusted geometric means (gMean). Standard deviation is actually Intra individual geometric coefficient variation (gCV)

11. Primary Outcome: C6hr of Deleobuvir Reduction Metabolite CD 6168
Description: Concentration of an analyte in plasma at 6 hours
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Group A | Group B
Number analyzed (Participants) | 16 | 19
nmol/L
  Day 9 (N=0, 17) | NA (NA) — Not calculated as this timepoint was not planned to be analysed for group A. | 2250 (137)
  Day 17 (N=14, 19) | 6980 (128) | 10200 (81.0)
  Day 66 (N=13, 14) | 3360 (139) | 7460 (123)
Statistical Analysis 1: Comparison: Group B; Day 17 vs. Day 9; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 1.0000, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 17 vs. Day 9 (%) = 450.51, 90% CI 2-sided [343.67 to 590.57], Standard Deviation 48.0 — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: Group B; Day 66 vs. Day 9; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 0.9996, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 66 vs. Day 9 (%) = 341.96, 90% CI 2-sided [229.22 to 510.13], Standard Deviation 61.1 — [estimate comment as in outcome 10, analysis 2]

12. Primary Outcome: AUC 0-6hr of Deleobuvir Reduction Metabolite CD 6168
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to 6 hours
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | Group A | Group B
Number analyzed (Participants) | 16 | 19
nmol*h/L
  Day 9 (N=0, 17) | NA (NA) — Not calculated as this timepoint was not planned to be analysed for group A. | 13300 (123)
  Day 17 (N=14, 19) | 41700 (130) | 62200 (82.7)
  Day 66 (N=13, 15) | 19300 (134) | 39100 (133)
Statistical Analysis 1: Comparison: Group B; Day 17 vs. Day 9; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 1.0000, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 17 vs. Day 9 (%) = 466.92, 90% CI 2-sided [357.02 to 610.66], Standard Deviation 47.6 — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: Group B; Day 66 vs. Day 9; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 0.9972, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 66 vs. Day 9 (%) = 298.57, 90% CI 2-sided [187.22 to 476.15], Standard Deviation 79.2 — [estimate comment as in outcome 10, analysis 2]

13. Primary Outcome: Cmax of Deleobuvir Metabolite CD 6168 ag (Acylglucuronide)
Description: Maximum concentration of an analyte in plasma
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Group A | Group B
Number analyzed (Participants) | 16 | 19
nmol/L
  Day 9 (N=0, 17) | NA (NA) — Not calculated as this timepoint was not planned to be analysed for group A. | 203 (135)
  Day 17 (N=14, 19) | 596 (143) | 1130 (115)
  Day 66 (N=13, 15) | 386 (111) | 806 (125)
Statistical Analysis 1: Comparison: Group B; Day 17 vs. Day 9; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 1.0000, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 17 vs. Day 9 (%) = 528.95, 90% CI 2-sided [415.88 to 672.75], Standard Deviation 42.0 — Relative bioavailability of BI CD 6168-ag at Day 17 vs. Day 9 -was estimated by the ratios of the adjusted geometric means (gMean). Standard deviation is actually Intra individual geometric coefficient variation (gCV)
Statistical Analysis 2: Comparison: Group B; Day 66 vs. Day 9; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 0.9998, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 66 vs. Day 9 (%) = 384.00, 90% CI 2-sided [251.56 to 586.16], Standard Deviation 69.2 — Relative bioavailability of BI CD 6168-ag at Day 66 vs. Day 9 -was estimated by the ratios of the adjusted geometric means (gMean). Standard deviation is actually Intra individual geometric coefficient variation (gCV)

14. Primary Outcome: C6hr of Deleobuvir Metabolite CD 6168 ag (Acylglucuronide)
Description: Concentration of an analyte in plasma at 6 hours
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Group A | Group B
Number analyzed (Participants) | 16 | 19
nmol/L
  Day 9 (N=0, 17) | NA (NA) — Not calculated as this timepoint was not planned to be analysed for group A. | 159 (165)
  Day 17 (N=14, 19) | 508 (138) | 962 (117)
  Day 66 (N=13, 14) | 295 (128) | 712 (143)
Statistical Analysis 1: Comparison: Group B; Day 17 vs. Day 9; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 1.0000, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 17 vs. Day 9 (%) = 569.81, 90% CI 2-sided [447.49 to 725.57], Standard Deviation 42.2 — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 2: Comparison: Group B; Day 66 vs. Day 9; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 0.9999, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 66 vs. Day 9 (%) = 441.89, 90% CI 2-sided [286.81 to 680.82], Standard Deviation 66.9 — [estimate comment as in outcome 13, analysis 2]

15. Primary Outcome: AUC 0-6hr of Deleobuvir Metabolite CD 6168 ag (Acylglucuronide)
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to 6 hours
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | Group A | Group B
Number analyzed (Participants) | 16 | 19
nmol*h/L
  Day 9 (N=0, 17) | NA (NA) — Not calculated as this timepoint was not planned to be analysed for group A. | 893 (142)
  Day 17 (N=14, 19) | 2980 (151) | 5700 (123)
  Day 66 (N=13, 15) | 1620 (133) | 3510 (143)
Statistical Analysis 1: Comparison: Group B; Day 17 vs. Day 9; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 1.0000, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 17 vs. Day 9 (%) = 606.29, 90% CI 2-sided [471.42 to 779.74], Standard Deviation 44.2 — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 2: Comparison: Group B; Day 66 vs. Day 9; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 0.9994, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 66 vs. Day 9 (%) = 377.98, 90% CI 2-sided [233.48 to 611.91], Standard Deviation 82.0 — [estimate comment as in outcome 13, analysis 2]

16. Primary Outcome: Cmax of Caffeine
Description: Maximum concentration of an analyte in plasma
Time Frame: 5 min before and 1 hour (h), 2h, 3h, 4h, 5h, 6h, 8h, 10h, 11:55h, 15h, 23:55h, 26h, 28h, 29:55h, 32h after first drug administration on day 1 also 5 min before, 1h, 2h, 3h, 4h, 5h, 5:55h, 8h, 10h, 11:55h, 15h, 23:55h after drug on days 9, 17 and 66.
Population: PKS. This endpoint was not planned to be analysed for groups C, D and E
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Group A | Group B
Number analyzed (Participants) | 16 | 19
ng/mL
  Day 1 (N=16, 19) | 5170 (46.2) | 5340 (38.2)
  Day 9 (N=15, 17) | 4890 (57.7) | 7220 (37.1)
  Day 17 (N=14, 19) | 4830 (47.5) | 6530 (52.3)
  Day 66 (N=13, 15) | 5590 (49.6) | 6450 (32.4)
Statistical Analysis 1: Comparison: Group A; Day 9 vs. Day 1; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 0.0500, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 9 vs. Day 1 (%) = 97.03, 90% CI 2-sided [80.00 to 117.69], Standard Deviation 30.8 — Relative bioavailability of caffeine at Day 9 vs. Day 1 -was estimated by the ratios of the adjusted geometric means (gMean). Standard deviation is actually Intra individual geometric coefficient variation (gCV)
Statistical Analysis 2: Comparison: Group A; Day 17 vs. Day 1; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 0.0564, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 17 vs. Day 1 (%) = 97.10, 90% CI 2-sided [79.37 to 118.79], Standard Deviation 31.2 — Relative bioavailability of caffeine at Day 17 vs. Day 1 -was estimated by the ratios of the adjusted geometric means (gMean). Standard deviation is actually Intra individual geometric coefficient variation (gCV)
Statistical Analysis 3: Comparison: Group A; Day 66 vs. Day 1; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 0.2375, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 66 vs. Day 1 (%) = 114.38, 90% CI 2-sided [92.36 to 141.66], Standard Deviation 31.9 — Relative bioavailability of caffeine at Day 66 vs. Day 1 -was estimated by the ratios of the adjusted geometric means (gMean). Standard deviation is actually Intra individual geometric coefficient variation (gCV)
Statistical Analysis 4: Comparison: Group B; Day 9 vs. Day 1; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 0.9082, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 9 vs. Day 1 (%) = 139.07, 90% CI 2-sided [121.63 to 159.00], Standard Deviation 22.8 — [estimate comment as in outcome 16, analysis 1]
Statistical Analysis 5: Comparison: Group B; Day 17 vs. Day 1; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 0.4111, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 17 vs. Day 1 (%) = 122.37, 90% CI 2-sided [104.11 to 143.84], Standard Deviation 29.3 — [estimate comment as in outcome 16, analysis 2]
Statistical Analysis 6: Comparison: Group B; Day 66 vs. Day 1; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 0.3719, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 66 vs. Day 1 (%) = 121.43, 90% CI 2-sided [104.24 to 141.45], Standard Deviation 24.7 — [estimate comment as in outcome 16, analysis 3]

17. Primary Outcome: AUC 0-infinity of Caffeine
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity.
Time Frame: as for outcome 16
Population: PKS. This endpoint was not planned to be analysed for groups C, D and E
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Group A | Group B
Number analyzed (Participants) | 16 | 19
ng*h/mL
  Day 1 (N=16, 19) | 54900 (130) | 77500 (119)
  Day 9 (N=15, 15) | 42100 (96) | 142000 (109)
  Day 17 (N=14, 19) | 71900 (169) | 170000 (203)
  Day 66 (N=13, 15) | 120000 (220) | 159000 (138)
Statistical Analysis 1: Comparison: Group A; Day 9 vs. Day 1; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 0.1037, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 9 vs. Day 1 (%) = 88.37, 90% CI 2-sided [77.39 to 100.89], Standard Deviation 20.8 — [estimate comment as in outcome 16, analysis 1]
Statistical Analysis 2: Comparison: Group A; Day 17 vs. Day 1; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 0.8723, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 17 vs. Day 1 (%) = 159.11, 90% CI 2-sided [111.06 to 227.93], Standard Deviation 57.8 — [estimate comment as in outcome 16, analysis 2]
Statistical Analysis 3: Comparison: Group A; Day 66 vs. Day 1; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 0.9830, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 66 vs. Day 1 (%) = 259.57, 90% CI 2-sided [150.65 to 447.21], Standard Deviation 92.5 — [estimate comment as in outcome 16, analysis 3]
Statistical Analysis 4: Comparison: Group B; Day 9 vs. Day 1; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 0.9689, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 9 vs. Day 1 (%) = 163.95, 90% CI 2-sided [129.52 to 207.52], Standard Deviation 38.1 — [estimate comment as in outcome 16, analysis 1]
Statistical Analysis 5: Comparison: Group B; Day 17 vs. Day 1; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 0.9933, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 17 vs. Day 1 (%) = 219.88, 90% CI 2-sided [153.84 to 314.26], Standard Deviation 70.4 — [estimate comment as in outcome 16, analysis 2]
Statistical Analysis 6: Comparison: Group B; Day 66 vs. Day 1; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 0.9865, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 66 vs. Day 1 (%) = 214.40, 90% CI 2-sided [145.88 to 315.09], Standard Deviation 66.8 — [estimate comment as in outcome 16, analysis 3]

18. Primary Outcome: Cmax of Tolbutamide
Description: Maximum concentration of an analyte in plasma
Time Frame: as for outcome 16
Population: PKS. This endpoint was not planned to be analysed for groups C, D and E
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Group A | Group B
Number analyzed (Participants) | 16 | 19
nmol/L
  Day 1 (N=16, 19) | 152000 (30.8) | 170000 (18.6)
  Day 9 (N=15, 17) | 146000 (28.1) | 158000 (22.8)
  Day 17 (N=14, 19) | 130000 (24.7) | 126000 (32.0)
  Day 66 (N=13, 15) | 110000 (32.3) | 127000 (25.0)
Statistical Analysis 1: Comparison: Group A; Day 9 vs. Day 1; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 0.0015, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 9 vs. Day 1 (%) = 96.06, 90% CI 2-sided [87.77 to 105.13], Standard Deviation 14.2 — Relative bioavailability of tolbutamide at Day 9 vs. Day 1 -was estimated by the ratios of the adjusted geometric means (gMean). Standard deviation is actually Intra individual geometric coefficient variation (gCV)
Statistical Analysis 2: Comparison: Group A; Day 17 vs. Day 1; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 0.1617, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 17 vs. Day 1 (%) = 85.41, 90% CI 2-sided [76.32 to 95.57], Standard Deviation 17.2 — Relative bioavailability of tolbutamide at Day 17 vs. Day 1 -was estimated by the ratios of the adjusted geometric means (gMean). Standard deviation is actually Intra individual geometric coefficient variation (gCV)
Statistical Analysis 3: Comparison: Group A; Day 66 vs. Day 1; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 0.8930, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 66 vs. Day 1 (%) = 73.26, 90% CI 2-sided [65.03 to 82.54], Standard Deviation 17.5 — Relative bioavailability of tolbutamide at Day 66 vs. Day 1 -was estimated by the ratios of the adjusted geometric means (gMean). Standard deviation is actually Intra individual geometric coefficient variation (gCV)
Statistical Analysis 4: Comparison: Group B; Day 9 vs. Day 1; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 0.0005, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 9 vs. Day 1 (%) = 92.23, 90% CI 2-sided [86.67 to 98.13], Standard Deviation 10.5 — [estimate comment as in outcome 18, analysis 1]
Statistical Analysis 5: Comparison: Group B; Day 17 vs. Day 1; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 0.8646, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 17 vs. Day 1 (%) = 73.93, 90% CI 2-sided [65.55 to 83.39], Standard Deviation 21.6 — [estimate comment as in outcome 18, analysis 2]
Statistical Analysis 6: Comparison: Group B; Day 66 vs. Day 1; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 0.8378, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 66 vs. Day 1 (%) = 75.42, 90% CI 2-sided [68.15 to 83.45], Standard Deviation 16.4 — [estimate comment as in outcome 18, analysis 3]

19. Primary Outcome: AUC 0-infinity of Tolbutamide
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity.
Time Frame: as for outcome 16
Population: PKS. This endpoint was not planned to be analysed for groups C, D and E
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | Group A | Group B
Number analyzed (Participants) | 16 | 19
nmol*h/L
  Day 1 (N=16, 19) | 1940000 (42.5) | 2220000 (29.4)
  Day 9 (N=13, 17) | 1800000 (41.3) | 1940000 (36.5)
  Day 17 (N=14, 18) | 1520000 (36.4) | 1410000 (27.9)
  Day 66 (N=12, 15) | 1330000 (40.1) | 1390000 (33.2)
Statistical Analysis 1: Comparison: Group A; Day 9 vs. Day 1; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 0.0005, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 9 vs. Day 1 (%) = 98.17, 90% CI 2-sided [90.15 to 106.91], Standard Deviation 12.3 — [estimate comment as in outcome 18, analysis 1]
Statistical Analysis 2: Comparison: Group A; Day 17 vs. Day 1; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 0.3638, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 17 vs. Day 1 (%) = 81.26, 90% CI 2-sided [75.19 to 87.82], Standard Deviation 11.7 — [estimate comment as in outcome 18, analysis 2]
Statistical Analysis 3: Comparison: Group A; Day 66 vs. Day 1; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 0.8975, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 66 vs. Day 1 (%) = 70.93, 90% CI 2-sided [60.44 to 83.22], Standard Deviation 22.6 — [estimate comment as in outcome 18, analysis 3]
Statistical Analysis 4: Comparison: Group B; Day 9 vs. Day 1; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 0.1144, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 9 vs. Day 1 (%) = 86.37, 90% CI 2-sided [77.62 to 96.11], Standard Deviation 18.1 — [estimate comment as in outcome 18, analysis 1]
Statistical Analysis 5: Comparison: Group B; Day 17 vs. Day 1; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 1.0000, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 17 vs. Day 1 (%) = 64.66, 90% CI 2-sided [60.42 to 69.20], Standard Deviation 11.8 — [estimate comment as in outcome 18, analysis 2]
Statistical Analysis 6: Comparison: Group B; Day 66 vs. Day 1; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 0.9988, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 66 vs. Day 1 (%) = 63.75, 90% CI 2-sided [57.19 to 71.07], Standard Deviation 17.3 — [estimate comment as in outcome 18, analysis 3]

20. Primary Outcome: Cmax of Midazolam
Description: Maximum concentration of an analyte in plasma
Time Frame: as for outcome 16
Population: PKS. This endpoint was not planned to be analysed for groups C, D and E
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Group A | Group B
Number analyzed (Participants) | 16 | 19
nmol/L
  Day 1 (N=16, 19) | 21.1 (38.3) | 23.8 (41.2)
  Day 9 (N=15, 17) | 29.9 (34.7) | 29.8 (44.3)
  Day 17 (N=14, 19) | 31.9 (36.6) | 28.8 (46.9)
  Day 66 (N=13, 15) | 21.3 (34.0) | 23.2 (40.4)
Statistical Analysis 1: Comparison: Group A; Day 9 vs. Day 1; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 0.9749, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 9 vs. Day 1 (%) = 144.78, 90% CI 2-sided [128.30 to 163.36], Standard Deviation 19.0 — Relative bioavailability of Midazolam at Day 9 vs. Day 1 -was estimated by the ratios of the adjusted geometric means (gMean). Standard deviation is actually Intra individual geometric coefficient variation (gCV)
Statistical Analysis 2: Comparison: Group A; Day 17 vs. Day 1; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 0.9703, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 17 vs. Day 1 (%) = 152.94, 90% CI 2-sided [128.60 to 181.89], Standard Deviation 26.8 — Relative bioavailability of Midazolam at Day 17 vs. Day 1 -was estimated by the ratios of the adjusted geometric means (gMean). Standard deviation is actually Intra individual geometric coefficient variation (gCV)
Statistical Analysis 3: Comparison: Group A; Day 66 vs. Day 1; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 0.0500, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 66 vs. Day 1 (%) = 102.99, 90% CI 2-sided [84.85 to 124.99], Standard Deviation 29.3 — Relative bioavailability of Midazolam at Day 66 vs. Day 1 -was estimated by the ratios of the adjusted geometric means (gMean). Standard deviation is actually Intra individual geometric coefficient variation (gCV)
Statistical Analysis 4: Comparison: Group B; Day 9 vs. Day 1; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 0.4697, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 9 vs. Day 1 (%) = 124.22, 90% CI 2-sided [107.91 to 142.99], Standard Deviation 24.1 — [estimate comment as in outcome 20, analysis 1]
Statistical Analysis 5: Comparison: Group B; Day 17 vs. Day 1; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 0.2906, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 17 vs. Day 1 (%) = 120.74, 90% CI 2-sided [108.47 to 134.38], Standard Deviation 19.2 — [estimate comment as in outcome 20, analysis 2]
Statistical Analysis 6: Comparison: Group B; Day 66 vs. Day 1; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 0.0460, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 66 vs. Day 1 (%) = 93.95, 90% CI 2-sided [80.33 to 109.86], Standard Deviation 25.2 — [estimate comment as in outcome 20, analysis 3]

21. Primary Outcome: AUC 0-infinity of Midazolam
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity.
Time Frame: as for outcome 16
Population: PKS. This endpoint was not planned to be analysed for groups C, D and E
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | Group A | Group B
Number analyzed (Participants) | 16 | 19
nmol*h/L
  Day 1 (N=16, 19) | 79.7 (59.1) | 107 (40.7)
  Day 9 (N=15, 17) | 117 (58.2) | 130 (66.9)
  Day 17 (N=14, 19) | 127 (50.2) | 140 (51.8)
  Day 66 (N=13, 15) | 75.5 (46.7) | 95.6 (41.6)
Statistical Analysis 1: Comparison: Group A; Day 9 vs. Day 1; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 0.9941, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 9 vs. Day 1 (%) = 151.66, 90% CI 2-sided [134.79 to 170.64], Standard Deviation 18.5 — [estimate comment as in outcome 20, analysis 1]
Statistical Analysis 2: Comparison: Group A; Day 17 vs. Day 1; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 0.9926, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 17 vs. Day 1 (%) = 163.42, 90% CI 2-sided [137.91 to 193.64], Standard Deviation 26.0 — [estimate comment as in outcome 20, analysis 2]
Statistical Analysis 3: Comparison: Group A; Day 66 vs. Day 1; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 0.0392, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 66 vs. Day 1 (%) = 98.14, 90% CI 2-sided [81.20 to 118.63], Standard Deviation 28.1 — [estimate comment as in outcome 20, analysis 3]
Statistical Analysis 4: Comparison: Group B; Day 9 vs. Day 1; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 0.4374, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 9 vs. Day 1 (%) = 122.58, 90% CI 2-sided [99.15 to 151.55], Standard Deviation 37.2 — [estimate comment as in outcome 20, analysis 1]
Statistical Analysis 5: Comparison: Group B; Day 17 vs. Day 1; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 0.6470, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 17 vs. Day 1 (%) = 130.44, 90% CI 2-sided [107.57 to 158.18], Standard Deviation 35.3 — [estimate comment as in outcome 20, analysis 2]
Statistical Analysis 6: Comparison: Group B; Day 66 vs. Day 1; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 0.2372, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 66 vs. Day 1 (%) = 87.77, 90% CI 2-sided [70.32 to 109.54], Standard Deviation 36.9 — [estimate comment as in outcome 20, analysis 3]

22. Primary Outcome: Cmax of 1-OH-Midazolam (1-hydroxy-midazolam)
Description: Maximum concentration of an analyte in plasma
Time Frame: as for outcome 16
Population: PKS. This endpoint was not planned to be analysed for groups C, D and E
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Group A | Group B
Number analyzed (Participants) | 16 | 19
nmol/L
  Day 1 (N=16, 19) | 5.57 (36.4) | 6.68 (67.1)
  Day 9 (N=15, 17) | 6.50 (46.3) | 6.52 (46.9)
  Day 17 (N=14, 19) | 6.46 (42.7) | 5.02 (50.5)
  Day 66 (N=13, 15) | 5.05 (45.6) | 4.67 (45.2)
Statistical Analysis 1: Comparison: Group A; Day 9 vs. Day 1; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 0.1519, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 9 vs. Day 1 (%) = 117.67, 90% CI 2-sided [106.49 to 130.00], Standard Deviation 15.6 — Relative bioavailability of 1-OH-Midazolam at Day 9 vs. Day 1 -was estimated by the ratios of the adjusted geometric means (gMean). Standard deviation is actually Intra individual geometric coefficient variation (gCV)
Statistical Analysis 2: Comparison: Group A; Day17 vs. Day 1; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 0.2827, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 17 vs. Day 1 (%) = 117.01, 90% CI 2-sided [96.06 to 142.52], Standard Deviation 30.9 — Relative bioavailability of 1-OH-Midazolam at Day 17 vs. Day 1 -was estimated by the ratios of the adjusted geometric means (gMean). Standard deviation is actually Intra individual geometric coefficient variation (gCV)
Statistical Analysis 3: Comparison: Group A; Day 66 vs. Day 1; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 0.1326, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 66 vs. Day 1 (%) = 92.11, 90% CI 2-sided [74.38 to 114.07], Standard Deviation 32.6 — Relative bioavailability of 1-OH-Midazolam at Day 66 vs. Day 1 -was estimated by the ratios of the adjusted geometric means (gMean). Standard deviation is actually Intra individual geometric coefficient variation (gCV)
Statistical Analysis 4: Comparison: Group B; Day 9 vs. Day 1; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 0.0432, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 9 vs. Day 1 (%) = 95.55, 90% CI 2-sided [80.63 to 113.24], Standard Deviation 29.2 — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 5: Comparison: Group B; Day 17 vs. Day 1; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 0.7367, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 17 vs. Day 1 (%) = 75.19, 90% CI 2-sided [63.64 to 88.82], Standard Deviation 30.3 — [estimate comment as in outcome 22, analysis 2]
Statistical Analysis 6: Comparison: Group B; Day 66 vs. Day 1; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 0.8547, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 66 vs. Day 1 (%) = 70.14, 90% CI 2-sided [56.84 to 86.56], Standard Deviation 34.3 — [estimate comment as in outcome 22, analysis 3]

23. Primary Outcome: AUC 0-infinity of 1-OH-Midazolam (1-hydroxy-midazolam)
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity.
Time Frame: as for outcome 16
Population: PKS. This endpoint was not planned to be analysed for groups C, D and E
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | Group A | Group B
Number analyzed (Participants) | 16 | 19
nmol*h/L
  Day 1 (N=16, 19) | 23.6 (59.8) | 26.0 (65.2)
  Day 9 (N=15, 17) | 24.2 (35.9) | 28.5 (63.9)
  Day 17 (N=14, 19) | 23.5 (37.4) | 22.8 (49.8)
  Day 66 (N=13, 13) | 18.3 (26.7) | 20.8 (46.1)
Statistical Analysis 1: Comparison: Group A; Day 9 vs. Day 1; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 0.1159, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 9 vs. Day 1 (%) = 102.70, 90% CI 2-sided [77.89 to 135.39], Standard Deviation 45.9 — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 2: Comparison: Group A; Day 17 vs. Day 1; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 0.0651, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 17 vs. Day 1 (%) = 99.99, 90% CI 2-sided [78.33 to 127.64], Standard Deviation 38.7 — [estimate comment as in outcome 22, analysis 2]
Statistical Analysis 3: Comparison: Group A; Day 66 vs. Day 1; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 0.5658, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 66 vs. Day 1 (%) = 78.29, 90% CI 2-sided [62.50 to 98.07], Standard Deviation 34.3 — [estimate comment as in outcome 22, analysis 3]
Statistical Analysis 4: Comparison: Group B; Day 9 vs. Day 1; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 0.1286, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 9 vs. Day 1 (%) = 108.25, 90% CI 2-sided [87.46 to 133.99], Standard Deviation 37.2 — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 5: Comparison: Group B; Day 17 vs. Day 1; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 0.1898, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 17 vs. Day 1 (%) = 87.59, 90% CI 2-sided [73.56 to 104.30], Standard Deviation 31.8 — [estimate comment as in outcome 22, analysis 2]
Statistical Analysis 6: Comparison: Group B; Day 66 vs. Day 1; Test type: Non-Inferiority or Equivalence — p-value for ratio outside 80% to 125%; p = 0.5575, ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of gmeans Day 66 vs. Day 1 (%) = 78.42, 90% CI 2-sided [61.81 to 99.51], Standard Deviation 36.3 — [estimate comment as in outcome 22, analysis 3]

24. Primary Outcome: Cmax of Tenofovir
Description: Maximum concentration of an analyte in plasma.
Time Frame: PK plasma samples were taken at: 5 minutes before drug administration and 1 hour (h), 2h, 3h, 4h, 5h, 5:55h, 8h, 10h, 11:55h, 15h, 23:55h after first drug administration on days 9 and 17
Population: PKS. Due to Boehringer Ingelheim's decision not to pursue the development of this substance, the extent of the statistical analysis was limited to selected endpoints. No further analysis is planned for the endpoints which were not related to patient efficacy or safety.
Arm/Group | Group C
Number analyzed (Participants) | 0

25. Primary Outcome: C24hr of Tenofovir
Description: Concentration of an analyte in plasma at 24 hours.
Time Frame: as for outcome 24
Population: as for outcome 24
Arm/Group | Group C
Number analyzed (Participants) | 0

26. Primary Outcome: AUC 0-24hr of Tenofovir
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to 24 hours.
Time Frame: as for outcome 24
Population: as for outcome 24
Arm/Group | Group C
Number analyzed (Participants) | 0

27. Primary Outcome: Cmax of Raltegravir
Description: Maximum concentration of an analyte in plasma.
Time Frame: as for outcome 24
Population: as for outcome 24
Arm/Group | Group E
Number analyzed (Participants) | 0

28. Primary Outcome: C12hr of Raltegravir
Description: Concentration of an analyte in plasma at 12 hours.
Time Frame: as for outcome 24
Population: as for outcome 24
Arm/Group | Group E
Number analyzed (Participants) | 0

29. Primary Outcome: AUC 0-12hr of Raltegravir
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to 12 hours.
Time Frame: as for outcome 24
Population: as for outcome 24
Arm/Group | Group E
Number analyzed (Participants) | 0

30. Secondary Outcome: Number of Participants With Sustained Virological Response (SVR12)
Description: Sustained virologic response (SVR12): Plasma Hepatitis C virus Ribonucleic acid (HCV RNA) level <25 IU/mL(international units per millilitre) undetectable at 12 weeks after the end of treatment. SVR12 was analyzed in a descriptive manner using frequency of participants who achieved SVR12.
Time Frame: 12 weeks post treatment
Population: Treated set (TRT): This subject set includes all patients who were dispensed trial medication and were documented to have taken at least one dose of trial drug.
Measure: Number; unit: Participants
Arm/Group | Group A | Group B | Group C | Group D | Group E
Number analyzed (Participants) | 16 | 19 | 16 | 14 | 7
Participants | 13 | 13 | 11 | 10 | 3

ADVERSE EVENTS:
Time Frame: From first drug administration until last drug administration plus 28 days, up to 28 weeks.
Arm/Group | Group A | Group B | Group C | Group D | Group E
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/19 | 1/16 | 2/14 | 0/7
Other Adverse Events (participants affected / at risk) | 16/16 | 19/19 | 16/16 | 14/14 | 5/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A (N=16) | Group B (N=19) | Group C (N=16) | Group D (N=14) | Group E (N=7)
Colitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Complex partial seizures (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Acute psychosis (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Reactive psychosis (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group A (N=16) | Group B (N=19) | Group C (N=16) | Group D (N=14) | Group E (N=7)
Anaemia (Blood and lymphatic system disorders) | 1 | 3 | 3 | 1 | 2
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 2 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Cardiovascular disorder (Cardiac disorders) | 0 | 0 | 1 | 0 | 2
Palpitations (Cardiac disorders) | 3 | 0 | 1 | 1 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 2 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 1
Blepharospasm (Eye disorders) | 1 | 0 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 1 | 0 | 0 | 0 | 0
Eye irritation (Eye disorders) | 0 | 0 | 0 | 1 | 0
Eye pain (Eye disorders) | 2 | 0 | 0 | 0 | 0
Eyelids pruritus (Eye disorders) | 0 | 0 | 1 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 1 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 1 | 0 | 0
Ocular icterus (Eye disorders) | 1 | 3 | 2 | 5 | 1
Periorbital oedema (Eye disorders) | 0 | 1 | 0 | 0 | 0
Photophobia (Eye disorders) | 1 | 0 | 0 | 0 | 0
Retinal exudates (Eye disorders) | 0 | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 3 | 1 | 0 | 0
Visual acuity reduced (Eye disorders) | 1 | 0 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 3 | 2 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 4 | 0 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 2 | 4 | 4 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 4 | 3 | 0
Abdominal rigidity (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Anal pruritus (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Anorectal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Chapped lips (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 3 | 4 | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 5 | 10 | 4 | 3 | 3
Dry mouth (Gastrointestinal disorders) | 4 | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 6 | 3 | 3 | 4 | 2
Faeces discoloured (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | 0
Gastrointestinal motility disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Lip dry (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Lip erosion (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Lip haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Lip oedema (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Lip pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Mucous stools (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 12 | 16 | 12 | 10 | 2
Oral discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Oral disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Paraesthesia oral (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Tongue discolouration (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 5 | 11 | 7 | 5 | 1
Asthenia (General disorders) | 0 | 6 | 1 | 1 | 0
Chest discomfort (General disorders) | 1 | 0 | 1 | 0 | 0
Chills (General disorders) | 6 | 7 | 1 | 0 | 1
Energy increased (General disorders) | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 9 | 11 | 8 | 8 | 2
Feeling hot (General disorders) | 0 | 0 | 0 | 1 | 1
Feeling of body temperature change (General disorders) | 0 | 0 | 0 | 1 | 0
Feeling of relaxation (General disorders) | 0 | 1 | 0 | 0 | 0
Influenza like illness (General disorders) | 3 | 3 | 0 | 0 | 1
Injection site bruising (General disorders) | 0 | 1 | 0 | 0 | 0
Injection site haematoma (General disorders) | 1 | 0 | 0 | 0 | 0
Injection site pain (General disorders) | 1 | 0 | 0 | 0 | 0
Injection site reaction (General disorders) | 0 | 1 | 0 | 0 | 0
Local swelling (General disorders) | 0 | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 3 | 0 | 0 | 0
Nodule (General disorders) | 1 | 0 | 0 | 0 | 0
Oedema (General disorders) | 0 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 1
Pain (General disorders) | 1 | 1 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 1 | 0 | 1 | 0
Pyrexia (General disorders) | 3 | 2 | 0 | 0 | 0
Temperature intolerance (General disorders) | 0 | 1 | 0 | 0 | 0
Tenderness (General disorders) | 0 | 1 | 0 | 0 | 0
Unevaluable event (General disorders) | 1 | 0 | 0 | 0 | 0
Vessel puncture site pain (General disorders) | 0 | 2 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 4 | 7 | 4
Jaundice (Hepatobiliary disorders) | 1 | 2 | 3 | 4 | 0
Body tinea (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 1 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Gastritis viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Genital herpes (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 3 | 0 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 2 | 3 | 2
Oral herpes (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Post procedural infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Tinea pedis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Scratch (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Skin wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Sunburn (Injury, poisoning and procedural complications) | 3 | 2 | 1 | 3 | 2
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 2 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1 | 0
Blood pressure increased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 1 | 0
Glomerular filtration rate decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 1 | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 6 | 8 | 3 | 5 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Food craving (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 4 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 1 | 0 | 1
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 4 | 3 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Burning sensation (Nervous system disorders) | 3 | 1 | 0 | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 1 | 1 | 1 | 1 | 0
Dizziness (Nervous system disorders) | 6 | 5 | 1 | 1 | 0
Dysaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 3 | 2 | 1 | 1 | 0
Headache (Nervous system disorders) | 9 | 9 | 5 | 5 | 1
Hyperaesthesia (Nervous system disorders) | 2 | 0 | 0 | 0 | 0
Hypertonia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 1 | 0 | 0 | 1
Hypogeusia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 2 | 0 | 0 | 0 | 0
Mental impairment (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 2 | 2 | 1 | 1
Parosmia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Psychomotor hyperactivity (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 1 | 1 | 0
Sleep phase rhythm disturbance (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Affect lability (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 2 | 2 | 0 | 1
Disorientation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Flat affect (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Frustration (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Hallucination, visual (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Impatience (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 8 | 5 | 3 | 0 | 0
Irritability (Psychiatric disorders) | 5 | 4 | 1 | 0 | 1
Libido increased (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 1 | 3 | 1
Stress (Psychiatric disorders) | 1 | 1 | 1 | 0 | 0
Chromaturia (Renal and urinary disorders) | 2 | 2 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 2 | 1 | 0 | 0 | 0
Renal disorder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 1 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 1 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2 | 1 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 3 | 0 | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 4 | 3 | 2 | 2
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 3 | 2 | 0 | 3 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 4 | 1 | 0 | 0
Macule (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Nail atrophy (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 3 | 6 | 3 | 0 | 2
Papule (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 9 | 8 | 2 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 10 | 6 | 9 | 2
Pruritus generalised (Skin and subcutaneous tissue disorders) | 2 | 2 | 1 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 6 | 7 | 5 | 0 | 4
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Skin reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3 | 0
Skin warm (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Vitiligo (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Xeroderma (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Tooth extraction (Surgical and medical procedures) | 0 | 2 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Hot flush (Vascular disorders) | 0 | 1 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 2 | 0
Pallor (Vascular disorders) | 0 | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
BI decided to stop the further development of the interferon-free combination therapy for Hepatitis C in December 2013 so the recruitment was stopped after 7 patients had entered Group E also PK analyses for Groups C to E were not performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.